CLINICAL TRIAL: NCT02200991
Title: A Randomized, Multicenter, Open-Label, Parallel-Group, 28 Days Phase IV Study Comparing The Postprandial Plasma Glucose Profile of Lixisenatide With That of Sitagliptin Add-On to Insulin Glargine in Type 2 Diabetes Mellitus
Brief Title: Effect of Lixisenatide on Postprandial Plasma Glucose Compared to Sitagliptin in Combination With Insulin Glargine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LIXISL06651; U1111-1159-5323 (UTN)
Record Dates: First submitted 2014-07-23; First posted 2014-07-25 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — lixisenatide; Sitagliptin Phosphate; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lixisenatide (Experimental): Lyxumia solostar: Initially started with 10 μg once-daily and increased up to 20 μg once daily (dose increased by 5 μg every week), subcutaneous injection in the abdomen, administered 30 minutes before breakfast. The period of administration is 4 weeks.
  Lantus solostar as base treatment: Subcutaneous injection in the abdomen.
  Interventions: Drug: LIXISENATIDE AVE0010; Drug: Insulin glargine HOE901
- Sitagliptin - Januvia (Active Comparator): 50 mg tablet, administered orally once-daily, 30 minutes before breakfast. The period of administration is 4 weeks.
  Lantus solostar as base treatment: Subcutaneous injection in the abdomen.
  Interventions: Drug: Sitagliptin; Drug: Insulin glargine HOE901

INTERVENTIONS:
Drug: LIXISENATIDE AVE0010 — Pharmaceutical form:solution Route of administration: subcutaneous
  Arms: Lixisenatide
Drug: Sitagliptin — Pharmaceutical form:tablet Route of administration: oral
  Other Names: Januvia
  Arms: Sitagliptin - Januvia
Drug: Insulin glargine HOE901 — Pharmaceutical form:solution Route of administration: subcutaneous
  Other Names: Lantus

SUMMARY:
Primary Objective:

To demonstrate significant reduction in postprandial plasma glucose (ΔAUC0:30-4:30h) after a standardized breakfast from baseline to Day 29.

Secondary Objectives:

To demonstrate:

* Changes from baseline to Day 29 in maximum postprandial plasma glucose excursion, C-peptide and glucagon levels after a standardized breakfast
* Delaying gastric emptying (13C-acetic acid breath test)
* Safety and tolerability

DETAILED DESCRIPTION:
The duration per patient could be minimum of 38 to 47 days depending on screening visit and post-treatment observation allowances.

13C-acetic acid breath test will be conducted only in investigational site which can be implemented (about 40 patients).

ELIGIBILITY:
Inclusion criteria:

* Type 2 diabetes mellitus, treated with Lantus±SU; ≥5-year after diagnosis
* Aged 20-75 years
* Hemoglobin A1C ≥7.0%-≤10.0%
* Fasting plasma glucose ≤180 mg/dL at screening
* Stable treatment (±20%) with Lantus for 3 months or more prior to screening.
* Sulfonylurea dose stable for 3 months or more prior to screening

Exclusion criteria:

* Type 1 diabetes mellitus
* Pregnancy or lactation
* Hypersensitivity to Lixisenatide
* Severely uncontrolled glycemic situation
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy, stomach/gastric surgery or inflammatory bowel disease
* History of metabolic acidosis, including diabetic ketoacidosis, within 1 year prior to screening
* History within the previous 6 months of myocardial infarction, stroke or heart failure requiring hospitalization or drug or alcohol abuse
* Uncontrolled/inadequately controlled hypertension at the time of screening, with a resting systolic blood pressure >180 mmHg or diastolic blood pressure >95 mmHg
* Amylase and/or lipase >3 times or aspartate aminotransferase (AST), alanine aminotransferase (ALT) or alkaline phosphatase (ALP) >2 times the upper limit of the normal laboratory range
* End-stage renal disease and/or dialysis and clinically relevant history of gastrointestinal disease

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in postprandial plasma glucose at Day 29 after a standardized breakfast | Day 29 after first intake of investigational product

SECONDARY OUTCOMES:
Change from baseline in maximum postprandial plasma glucose excursion at Day 29 after a standardized breakfast | Day 29 after first intake of investigational product
Change from baseline in plasma C-peptide levels at Day 29 after a standardized breakfast | Day 29 after first intake of investigational product
Change from baseline in glucagon levels at Day 29 after a standardized breakfast | Day 29 after first intake of investigational product
Change in gastric emptying half life (13C-acetic acid breath test) | Day 29 after first intake of investigational product
Proportion of patients with adverse events | Up to Day 33 from the first intake of investigational medicinal product

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (20):
- Japan (20):
  - Investigational Site Number 392-107, Atsugi-shi
  - Investigational Site Number 392-125, Chiyoda-ku
  - Investigational Site Number 392-121, Chuoh-ku
  - Investigational Site Number 392-102, Ichihara-shi
  - Investigational Site Number 392-103, Kawaguchi-shi
  - Investigational Site Number 392-114, Kitamoto-shi
  - Investigational Site Number 392-122, Kobe
  - Investigational Site Number 392-126, Kumamoto
  - Investigational Site Number 392-127, Kumamoto
  - Investigational Site Number 392-101, Kyoto
  - Investigational Site Number 392-106, Matsudo-shi
  - Investigational Site Number 392-124, Mitaka-shi
  - Investigational Site Number 392-108, Mito
  - Investigational Site Number 392-119, Nerima-ku
  - Investigational Site Number 392-117, Okayama
  - Investigational Site Number 392-111, Sagamihara-shi
  - Investigational Site Number 392-110, Sapporo
  - Investigational Site Number 392-116, Satsumasendai-shi
  - Investigational Site Number 392-105, Shizuoka
  - Investigational Site Number 392-118, Suita-shi

REFERENCES:
- [Derived] Yamada Y, Senda M, Naito Y, Tamura M, Watanabe D, Shuto Y, Urita Y. Reduction of postprandial glucose by lixisenatide vs sitagliptin treatment in Japanese patients with type 2 diabetes on background insulin glargine: A randomized phase IV study (NEXTAGE Study). Diabetes Obes Metab. 2017 Sep;19(9):1252-1259. doi: 10.1111/dom.12945. Epub 2017 Apr 27. PMID 28345162